CLINICAL TRIAL: NCT01350492
Title: Impact of Exercise Training on Pain and Brain Function in Gulf War Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPLD-004-10S
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: pain; brain imaging; exercise
MeSH Terms: conditions — Pain; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Resistance exercise training
  Interventions: Behavioral: Resistance Exercise Training
- Arm 2 (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Resistance Exercise Training — 16 weeks of resistance exercise training for the treatment of chronic muscle pain compared to wait-list control
  Arms: Arm 1

SUMMARY:
This study is intended to test the influence of weight training on physical symptoms, physical activity and brain structure and function in Gulf War Veterans with chronic widespread muscle pain.

DETAILED DESCRIPTION:
Musculoskeletal pain in soldiers who returned from the Persian Gulf War is a serious problem. Numerous studies have reported musculoskeletal pain as a primary symptom of sick Gulf Veterans (GVs), with ~100,000 Veterans (~15%) reporting unresolved pain affecting their social and professional lives. Pain and other symptoms are often disabling with 1 in 7 United States Veterans seeking care for war-related health concerns and ~12% receiving disability compensation. Thus, a significant number of military personnel are no longer able to perform their duties due to medically unexplained symptoms including pain, fatigue and cognitive problems. Importantly, recent evidence suggests that chronic pain complaints in most GVs have not resolved. Similar problems appear to be on the horizon for Veterans from Operations Enduring and Iraqi Freedom. Understanding the pathophysiological consequences of chronic muscle pain is important for better determining both the efficacy and mechanism of treatments aimed at decreasing debilitating symptoms and improving physical function among Veterans coping with chronic pain.

Given the dearth of experimental data in GVs with chronic musculoskeletal pain (CMP), we have patterned much of our research in GVs after our research in fibromyalgia (FM), a disorder with a primary symptom of muscle and joint pain in civilians. Our work and the work of others suggest that FM pain is produced and maintained by central nervous system (CNS) dysregulation of nociceptive and pain processes. Our work also suggests that phenomena similar to those observed in FM may be occurring in GVs with CMP. Like FM patients, GVs with CMP, 1) are more sensitive to experimental pain stimuli, 2) exhibit exaggerated pain responses following acute exercise, 3) experience more muscle pain during acute exercise and 4) show augmented brain responses to both painful and non-painful experimental stimuli. These data suggest that some of the same pathophysiological mechanisms involved in FM may be maintaining chronic widespread muscle pain in GVs. Critical unanswered questions include whether promising treatments for CMP in GVs can affect laboratory measures of pain sensitivity and pain regulation and whether these changes relate to clinical improvements. We intend to begin to answer these questions by examining perceptual and brain hemodynamic responses to standardized painful stimuli and documenting their relationships to clinical outcomes before, during and upon completion of a viable, novel treatment for CMP.

There are no known efficacious treatments for GVs suffering CMP. Efficacy studies are needed to begin determining effective treatments for our Veterans following their service of our country. In FM, exercise training (both aerobic and resistance modes) is widely recognized as one of the few consistently efficacious treatments, resulting in improved well-being, increased physical function and in some cases decreased pain. One large scale treatment trial of aerobic exercise in GVs with chronic multi-symptom illness showed only modest improvements in pain, fatigue and mental health. We believe this trial had several limitations that greatly attenuated the treatment's effectiveness; consequently, it is premature to discount exercise training as a treatment for GVs with CMP. Further, we propose a novel approach that employs progressive resistance exercise training (RET) to treat GVs with CMP, while obtaining objective measures of nociceptive function, brain white matter tract pathways and total physical activity.

In addition to exercise performed as part of a structured training program, physical activity behaviors are important determinants of physical and mental health. Greater total physical activity levels are associated with increased physical function, improved mental health, increased energy and decreased symptoms of chronic pain. To our knowledge, none of the exercise training trials in FM have actually measured the impact of the exercise training on physical activity behaviors during daytime hours outside the intervention. It is plausible that the adoption of a structured exercise training program reduces physical activities performed during the rest of the day, and that this change in total physical activity could affect health outcomes. Objective measurement of physical activity will allow us to determine whether RET increases, decreases or has no impact on total physical activity levels in GVs with CMP. This will allow us to begin to characterize sub-groups who benefit the most from RET (e.g. potentially those GVs that maintain or increase their extra-intervention physical activity). Thus, in addition to supervised RET, we will objectively measure total physical activity levels outside of the intervention using accelerometers before, during and following treatment.

In summary, we propose to determine the efficacy of RET for the treatment of CMP and associated symptoms in GVs. In addition, we will assess the influence of RET on total physical activity, pain sensitivity and regulation, and brain white matter tracts. By applying functional neuroimaging techniques in conjunction with pain psychophysics we will test how the brains of Veterans with CMP respond to sensory stimuli and whether these responses can be modified by exercise training. We plan to use blood oxygen level dependent (BOLD) and diffusion tensor imaging (DTI) methods to evaluate the function of brain regions involved in pain processing and control and the microstructural properties of white matter tract pathways that connect these regions. In addition, we will determine the influence of RET on extra-intervention physical activity behaviors, testing a critical and unanswered question - whether total physical activity levels change as a result of engaging in a RET program in patients with CMP. The primary goals of this project will be accomplished by comparing GVs with CMP assigned to either RET or wait-list control (WLC) in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the Persian Gulf War
* Chronic muscle pain

Exclusion Criteria:

* Regular participation in resistance exercise
* Color blindness
* Claustrophobia
* Medical conditions that could explain the Veteran's pain
* Use of exclusionary drugs 3 weeks prior to testing
* Major depressive disorder with melancholic features
* Substance abuse
* Schizophrenia
* Bipolar disorder

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dane B. Cook, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2013 and March 2018, participants were recruited through digital and print advertisements in area medical centers, presentations at Veteran Service Organizations and via a mailed letter targeting Veterans from a VA database search. The first participant was enrolled in June 2013 and the last participant was enrolled in March 2018.
Pre-assignment Details: Following phone screening, 119 participants were invited to participate. Of those, 77 were enrolled and underwent a more substantial screening process. 54 participants were randomly assigned to a group. The remaining 23 participants were not assigned to a group as they were ineligible (n=17) or declined to continue (n=6).
Groups:
- Resistance Exercise Training: Resistance Exercise Training: 16 weeks of resistance exercise training, performed twice weekly, for the treatment of chronic muscle pain.
- Waitlist Control: Waitlist Control: Individuals assigned to this condition were asked to maintain their usual routine while enrolled. Upon completion they were offered the opportunity to undertake the resistance training protocol.
Period: Intervention
Arm/Group | Resistance Exercise Training | Waitlist Control
Started | 28 | 26
6-week MRI Scan | 24 | 22
11-week MRI Scan | 23 | 21
Completed | 23 | 20
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 3 | 1
Period: Post Intervention Follow-Up
Arm/Group | Resistance Exercise Training | Waitlist Control
Started | 23 | 20
6-month MRI Scan | 20 | 20
Completed | 17 | 18
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 6 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistance Exercise Training | Waitlist Control | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.71 (7.20) | 50.19 (5.64) | 49.94 (6.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 21 | 22 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, not Hispanic | 25 | 20 | 45
  White Hispanic | 2 | 3 | 5
  Black, not Hispanic | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 26 | 54
Marital Status [Count of Participants; unit: Participants]
  Married | 15 | 21 | 36
  Divorced | 6 | 4 | 10
  Never married | 3 | 1 | 4
  Widowed | 0 | 0 | 0
  Separated | 2 | 0 | 2
  Living as married | 2 | 0 | 2
Education [Count of Participants; unit: Participants]
  Did not finish high school | 0 | 1 | 1
  High school graduate | 4 | 6 | 10
  Some college | 11 | 6 | 17
  College graduate (including associates degree) | 9 | 11 | 20
  Some post-graduate | 1 | 0 | 1
  Graduate degree | 3 | 2 | 5
Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — Self-report measure of 13 items, each scored on a 0-4 scale, with a max score of 52. The higher the score the more catastrophizing thoughts are present. Developed by Sullivan and colleagues (1995), the scale is intended to quantify negative cognitive and emotional responses to actual or anticipated pain (e.g., feelings of hopelessness).
  units on a scale | 11.79 (8.72) | 8.65 (7.98) | 10.28 (8.44)
State Trait Anxiety Inventory (STAI) - Y2 Form [Mean (Standard Deviation); unit: units on a scale] — Self-report measure of 20 items, each scored on a 1-4 scale, with a minimum score of 20 and a max score of 80. Higher scores indicate greater anxiety. Developed by Spielberger and colleagues (1983), the Y2 form of the scale is intended to quantify trait anxiety, or anxiety level as a personality characteristic, experienced by the respondent.
  units on a scale | 37.57 (9.94) | 36.00 (9.21) | 36.81 (9.54)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — Self-report measure of 21 items, each scored on a 0-3 scale, with a max score of 63. The higher the score the more depressive symptoms are present. Developed by Beck (1978), the scale is intended to quantify characteristic attitudes and symptoms of depression (e.g., loss of interest and/or enjoyment).
  units on a scale | 9.07 (6.85) | 6.73 (6.62) | 7.94 (6.78)
Physical Activity (Accelerometer) [Mean (Standard Deviation); unit: Counts per day] — Physical activity is measured via accelerometer. The measure is a unit-less average of the number of counts per day. The higher the count, the greater the amount and intensity of physical activity accumulated over course of the day. Values range from 30,000 (sedentary) to 800,000 (highly active). Population: Measures were considered valid if the participant wore the accelerometer for at least 10 hr/day for 4 days. In addition, one of those 4 days must have been a weekend day (i.e., Saturday or Sunday). The sample is limited to only those participants with a valid baseline measure.
  Counts per day
    number analyzed (Participants) | 24 | 21 | 45
    (all) | 236520 (114918) | 337629 (165554) | 283704 (148202)
Physical Activity (Self-report) [Mean (Standard Deviation); unit: MET-minutes/week] — Total weekly self-reported physical activity was quantified using the International Physical Activity Questionnaire (IPAQ). The outcome is expressed as the number of metabolic equivalent (MET) minutes per week. One MET is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min, so 1 minute spent at rest is equal to 1 MET-minute. Respondents are only asked to report on physical activity of a light intensity or greater (≥3 METs, e.g., briskly walking). Higher values equal greater amount/intensity of activity.
  MET-minutes/week | 4820 (6094) | 5848 (7410) | 5315 (6715)
Fractional anisotropy (FA) at the corpus callosum [Mean (Standard Deviation); unit: Scalar value b/w 0-1] — Fractional anisotropy (FA) is a scalar value between 0 and 1 that describes the degree of anisotropy of a diffusion process. In the case of brain white matter integrity, it gives us an indication of the tract integrity at a particular region within the brain. 0 would indicate flow is completely unrestricted (low integrity), 1 that all flow is in the same direction (high integrity). In this instance we are using the FA at the body of the corpus callosum as an indicator of overall brain white matter integrity.
  Scalar value b/w 0-1 | 0.528 (0.030) | 0.521 (0.031) | 0.524 (0.030)

OUTCOME MEASURES:

1. Primary Outcome: Short Form McGill Pain Questionnaire Visual Analog Scale (VAS).
Description: The Short Form McGill Pain Questionnaire VAS ranges from 0 (No pain) to 100 (Worst possible pain). The respondent was asked to report how bad their pain has been over the past week. A higher score indicates a greater severity of pain.
Time Frame: 6 weeks, 11 weeks, 17 weeks and 6 and 12 months post intervention.
Population: Intent to treat population (all participants assigned to either resistance exercise training or wait-list control). Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resistance Exercise Training | Waitlist Control
Number analyzed (Participants) | 28 | 26
units on a scale
  6 weeks | 29.82 (22.12) | 37.08 (25.92)
  11 weeks | 30.07 (22.37) | 31.46 (21.78)
  17 weeks | 30.68 (24.12) | 35.12 (24.05)
  6 months | 31.5 (22.31) | 34.31 (25.66)
  12 months | 31.68 (23.37) | 33.58 (26.12)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Waitlist Control; General multivariate regression models were used to estimate the time averaged difference in pain ratings and other symptom scores (continuous measurements) between the treatment and the control group. In order to achieve 90% power, at alpha equal to .05, with an effect size of .6 (minimum effect size of clinical importance) and with a correlation of .6 between measurements from each individual, we estimated the necessary sample size at 34 subjects per group; Test type: Superiority; p = 0.680, Multivariate regression — The threshold for statistical significance was p = 0.05; A Generalized Linear Model was employed with repeated measurements of pain ratings as the multivariate dependent variables and group as covariate; Wilks' Lambda = 0.939

2. Primary Outcome: Physical Component Score (PCS) From the Veterans Rand 36 Item Heath Survey (VR-36).
Description: The PCS is a composite summary score of items from the VR-36 related to physical health. Individual subscale scores are z transformed using US normative data, multiplied by a factor score coefficient, summed, and transformed to a T-score of a distribution (Mean = 50; Standard Deviation = 10). Higher scores represent better physical health.
Time Frame: 6 weeks, 11 weeks, 17 weeks and 6 and 12 months post intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale, T-score transformed
Arm/Group | Resistance Exercise Training | Waitlist Control
Number analyzed (Participants) | 28 | 26
units on a scale, T-score transformed
  6 weeks | 43.01 (5.17) | 44.53 (6.06)
  11 weeks | 41.82 (5.95) | 43.37 (6.68)
  17 weeks | 42.66 (5.60) | 42.92 (5.80)
  6 months | 43.03 (5.96) | 43.94 (7.07)
  12 months | 41.14 (5.85) | 42.99 (6.59)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.854, Mulitvariate regression — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Wilks' Lambda = 0.960

3. Primary Outcome: Patients' Global Impression of Change (PGIC).
Description: The PGIC is a 7-item, self-report scale indicating the degree to which a patient has experienced any change since starting treatment. Each respondent was asked to rate "...the change (if any) in activity limitations, symptoms, emotions, and overall quality of life." related to their pain since beginning treatment. Scores range from 1, "No change (or condition has got worse)" to 7, "A great deal better, and a considerable improvement that has made all the difference." A higher score indicates greater improvement.
Time Frame: 6 weeks, 11 weeks, 17 weeks and 6 and 12 months post intervention.
Population: Intent to treat population (all participants assigned to either resistance exercise training or wait-list control). Last observation carried forward (LOCF) imputation method. THE PGIC, however, was not administered until the 6-week in-person visit. So participants who were withdrawn or lost to follow up before the 6-week visit were not included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resistance Exercise Training | Waitlist Control
Number analyzed (Participants) | 24 | 22
units on a scale
  6 weeks | 3.58 (1.59) | 1.77 (1.02)
  11 weeks | 3.67 (1.52) | 2.00 (0.87)
  17 weeks | 3.88 (1.83) | 2.05 (0.95)
  6 months | 3.21 (2.00) | 2.18 (1.47)
  12 months | 2.71 (1.81) | 2.45 (1.47)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0002, Multivariate regression — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Physical Activity (Accelerometer)
Description: Physical activity is measured via accelerometer. The measure is a unit-less average of the number of counts per day. The higher the count, the greater the amount and intensity of physical activity accumulated over course of the day. Values range from 30,000 (sedentary) to 800,000 (highly active).
Time Frame: 6 weeks, 11 weeks, 17 weeks and 6 and 12 months post intervention.
Population: Intent to treat population (all participants assigned to either resistance exercise training or wait-list control). Last observation carried forward (LOCF) imputation method. Sample is limited to only those participants with a valid baseline measure.
Measure: Mean (Standard Deviation); unit: Counts per day
Arm/Group | Resistance Exercise Training | Waitlist Control
Number analyzed (Participants) | 24 | 21
Counts per day
  6 weeks | 261012 (131113) | 299872 (124379)
  11 weeks | 267376 (133327) | 321253 (121150)
  17 weeks | 285157 (181804) | 305315 (122002)
  6 months | 267067 (168249) | 295661 (126297)
  12 months | 252940 (144748) | 300769 (132518)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.41, Multivariate regression — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Wilks' Lambda = 0.857

5. Secondary Outcome: Physical Activity (Self-report)
Description: Total weekly self-reported physical activity was quantified using the International Physical Activity Questionnaire (IPAQ). The outcome is expressed as the number of metabolic equivalent (MET) minutes per week. One MET is defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml O2 per kg body weight x min, so 1 minute spent at rest is equal to 1 MET-minute. Respondents are only asked to report on physical activity of a light intensity or greater (≥3 METs, e.g., briskly walking). Higher values equal greater amount/intensity of activity.
Time Frame: 6 weeks, 11 weeks, 17 weeks and 6 and 12 months post intervention.
Measure: Mean (Standard Deviation); unit: MET-minutes/week
Arm/Group | Resistance Exercise Training | Waitlist Control
Number analyzed (Participants) | 28 | 26
MET-minutes/week
  6 weeks | 4535 (5948) | 6824 (7944)
  11 weeks | 5856 (5912) | 4978 (7601)
  17 weeks | 4629 (4280) | 6491 (9020)
  6 months | 4232 (3771) | 6273 (9161)
  12 months | 4492 (4739) | 6113 (8709)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.16, Multivariate regression — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Wilks' Lambda = 0.828

6. Secondary Outcome: Brain Structure: White Matter Tract Integrity, Operationalized With Fractional Anisotropy (FA) Measures at the Body of the Corpus Callosum.
Description: Fractional anisotropy (FA) is a scalar value between 0 and 1 that describes the degree of anisotropy of a diffusion process. In the case of brain white matter integrity, it gives us an indication of the tract integrity at a particular region within the brain. 0 would indicate flow is completely unrestricted (no integrity), 1 that all flow is in the same direction (high integrity). In this instance we are using the FA at the body of the corpus callosum as an indicator of overall brain white matter integrity.
Time Frame: 6 weeks, 11 weeks, 17 weeks and 6 and 12 months
Measure: Mean (Standard Deviation); unit: Scalar value b/w 0 and 1
Arm/Group | Resistance Exercise Training | Waitlist Control
Number analyzed (Participants) | 28 | 26
Scalar value b/w 0 and 1
  6 weeks | 0.5263 (0.0310) | 0.5213 (0.0325)
  11 weeks | 0.5256 (0.0312) | 0.5213 (0.0323)
  17 weeks | 0.5261 (0.0298) | 0.5224 (0.0313)
  6 months | 0.5262 (0.0303) | 0.5217 (0.0325)
  12 months | 0.5219 (0.0343) | 0.5203 (0.0329)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Waitlist Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.66, Multivariate regression — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 1, analysis 1]; Wilks' Lambda = 0.919

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Resistance Exercise Training | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 0/28 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT01350492/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT01350492/ICF_001.pdf